CLINICAL TRIAL: NCT01921270
Title: A Pilot Dose Ranging Study of Dysport® (AbobotulinumtoxinA) in the Treatment of Oromandibular Dystonia
Brief Title: Dysport for the Treatment of OMD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Principal Investigator, Stewart Factor, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00064292
Record Dates: First submitted 2013-08-09; First posted 2013-08-13 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Oral Dystonia; Tardive Dystonia
Keywords: Oromandibular Dystonia; Oral Dystonia; Tardive Dystonia; botulinum toxin; abobotulinumtoxinA
MeSH Terms: conditions — Tardive Dyskinesia | interventions — abobotulinumtoxinA

STUDY DESIGN:
Masking Description: Evaluators will review the videotaped examinations, presented in a random order, using the Global Dystonia Rating scale (GDS). The evaluators will rate the dystonia at baseline (injection visit) and 6 weeks after injection.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dysport Injections (Experimental): Participants with OMD who have been previously treated with any botulinum toxin Type A will be injected with Dysport®.
  Interventions: Drug: Low Dose - AbobotulinumtoxinA

INTERVENTIONS:
Drug: Low Dose - AbobotulinumtoxinA — Participants will receive low dose AbobotulinumtoxinA injections. Location of injections will be determined by the clinician to treat the individual's dystonic symptom.
  Muscles that may be included for in injection for OMD with Jaw Closing:
  Medial Pterygoid 50 units, Masseter 25 units
  Muscles that may be included in injection for OMD with Jaw Opening:
  Lateral Pterygoid 50 units, Anterior digastrics 10 units
  Muscle that will be included in injection for OMD with Tongue Protrusion:
  Genioglossus 7.5 units
  Other Names: Dysport

SUMMARY:
The purpose of this study is to study the efficacy and safety of AbobotulinumtoxinA (Dysport) for use in Oromandibular Dystonia (OMD).

DETAILED DESCRIPTION:
Oromandibular dystonia (OMD) is an uncommon, disabling form of cranial dystonia, involving involuntary movements of the lower facial, masticatory, and lingual muscles. This can cause jaw movements including opening, closure, protrusion, retraction, or deviation. Common additional facial movements involve grimacing or lip pursing. When there is tongue involvement, it usually presents as tongue protrusion or curling. Such patients are impaired in relation to eating, speaking and swallowing

This study aims to evaluate the efficacy and safety of a low dose of Dysport® deemed tolerable during phase 1 in subjects with oromandibular dystonia (OMD).

Participants will be injected with Dysport® only, with an unblinded open-label disclosure. The safety and efficacy pf receiving Dysport® will be recorded for all subjects that undergo injection. All subjects will be examined and videotaped at the injection visit, then at 6 and 12 weeks after injection with a standardized protocol. The primary outcome will be blinded examination scores of the videos performed after the study is complete.The evaluators will be three different movement disorders experts, not otherwise involved in the study, who will review the videotaped examinations, presented in a random order, using the Global Dystonia Rating scale (GDS). Evaluators will rate the dystonia at baseline (injection visit) and 6 weeks after injection.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of primary or tardive OMD
* moderate or severe severity, defined as GDS score ≥4 in either "lower face" or "jaw and tongue" section
* capability of attending the scheduled visits
* only those who have been previously injected with onabotulinumtoxinA and responded to that treatment, and are at least 12 weeks post last injection
* Women of childbearing age need to use contraception in order to be included.

Exclusion Criteria:

* Existence of a systemic disease that could confound the evaluation
* previous placement of Deep Brain Stimulation electrodes to treat dystonia
* concomitant oral medications that could interfere with the action of botulinum toxin Type A (e.g., aminoglycosides)
* on an unstable dosage of any medication prescribed to treat dystonia (e.g., benzodiazepines, baclofen or anticholinergics)
* any known hypersensitivity to any botulinum toxin preparation and allergy to cow's milk protein
* immunoresistance to other forms of botulinum toxin type A
* existence of a concomitant neuromuscular disorder (e.g., Myasthenia Gravis or Lambert-Eaton syndrome, etc)
* infection at the proposed injection sites
* pregnant women
* women of childbearing age NOT on contraception
* breastfeeding women
* inability to comply with scheduled visits
* patients who had been previously injected with botulinum toxin type A but who did not respond

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-08; Primary Completion 2017-02-08 (Actual); Study Completion 2017-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stewart A Factor, DO, Principal Investigator — Emory University
Locations (1):
- Wesley Woods Health Center; Emory University Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Background] Tan EK, Jankovic J. Botulinum toxin A in patients with oromandibular dystonia: long-term follow-up. Neurology. 1999 Dec 10;53(9):2102-7. doi: 10.1212/wnl.53.9.2102. PMID 10599789
- [Background] Rosales RL, Ng AR, Santos MM, Fernandez HH. The broadening application of chemodenervation in X-linked dystonia-parkinsonism (Part II): an open-label experience with botulinum toxin-A (Dysport(R)) injections for oromandibular, lingual, and truncal-axial dystonias. Int J Neurosci. 2011;121 Suppl 1:44-56. doi: 10.3109/00207454.2011.558260. PMID 21348790

RESULTS

PARTICIPANT FLOW:
Groups:
- Dysport Injections: Participants with OMD who have been previously treated with any botulinum toxin Type A were injected with Dysport®.
  Low Dose - AbobotulinumtoxinA: Participants will receive low dose AbobotulinumtoxinA injections. Location of injections will be determined by the clinician to treat the individual's dystonic symptom.
  Muscles that may be included for in injection for OMD with Jaw Closing:
  Medial Pterygoid 50 units, Masseter 25 units
  Muscles that may be included in injection for OMD with Jaw Opening:
  Lateral Pterygoid 50 units, Anterior digastrics 10 units
  Muscle that will be included in injection for OMD with Tongue Protrusion:
  Genioglossus 7.5 units
Period: Overall Study
Arm/Group | Dysport Injections
Started | 18
Completed | 17
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Participants who received low dose Dysport injections.
Arm/Group | Dysport Injections
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.83 (10.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Mean Global Dystonia Rating Scale Score as Measured by Blinded Rater
Description: This scale measures the severity of dystonia for the jaw and tongue by a blinded rater. Dystonia is rated from 0 to 10:
  0=No dystonia present, 1=Minimal dystonia, 5=Moderate dystonia,10=Most severe dystonia
Time Frame: Baseline, Week 6, Week 12
Population: Participants who received low dose Dysport injections and completed all study visits. Two participants received two injections each for which data from the second were included in the analysis. For change from baseline to week 6, 18 subjects analyzed, for change from baseline to week 12, 17 subjects analyzed as one subject dropped out at 6 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport Injections
Number analyzed (Participants) | 18
units on a scale
  Baseline | 3.80 (2.29)
  Week 6 | 3.57 (2.05)
  Week 12: number analyzed (Participants) | 17
  Week 12 | 3.71 (2.18)

2. Secondary Outcome: Change in Analogue Pain Scale Score
Description: Measure of jaw pain by visual analogue scale (0-100) where 0 represents "no pain" and 100 represents the "most severe pain".
Time Frame: Baseline, Week 12
Population: Data were not collected.
Arm/Group | Dysport Injections
Number analyzed (Participants) | 0

3. Secondary Outcome: Mean Sialorrhea Clinical Scale for Parkinson's Disease (SCS-PD) Score
Description: The SCS-PD measures drooling. Individual items are scored on a scale from 0-3 where 0 represents "never" and 3 represents "always". The overall maximum score is 21. A higher score indicates greater drooling severity. A lower score indicates lesser severity.
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport Injections
Number analyzed (Participants) | 18
units on a scale
  Baseline | 3.00 (3.91)
  Week 6 | 2.72 (4.28)
  Week 12: number analyzed (Participants) | 17
  Week 12 | 2.53 (3.20)

4. Secondary Outcome: Change in Number of Tongue Bites Per Day
Description: The patient will be asked to estimate how many times they tend to accidentally/involuntarily bite their tongue per day.
Time Frame: Baseline, Week 12
Population: Data were not collected.
Arm/Group | Dysport Injections
Number analyzed (Participants) | 0

5. Secondary Outcome: Mean Swallowing Disturbance Questionnaire (SDQ-20) Score
Description: Ease of chewing and swallowing will be assessed by the SDQ-20 (modified to exclude question 5 due to redundancy as it relates to drooling and question 15 which is not relevant to the study as it involves prior aspiration pneumonias). Individual items are scored from 0 (never) to 3 (very frequently). The overall score is the total for all items; a higher score indicating more frequent swallowing disturbance; a lower score indicating no or less frequent disturbance, with a possible maximum score of 39.
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport Injections
Number analyzed (Participants) | 18
units on a scale
  Baseline | 13.17 (9.51)
  Week 6 | 15.61 (8.56)
  Week 12: number analyzed (Participants) | 17
  Week 12 | 13.29 (8.54)

6. Secondary Outcome: Mean Fahn-Marsden Part B "Speech" Question (BFM-q21) Rating
Description: The Fahn-Marsden Part B "Speech" Question assesses the ease of producing speech. Responses range from 0=Normal, 1=Slightly involved, easily understood, 2=Some difficulty understanding, 3=Marked difficulty understanding.
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport Injections
Number analyzed (Participants) | 18
units on a scale
  Baseline | 1.33 (.91)
  Week 6 | .94 (.87)
  Week 12: number analyzed (Participants) | 17
  Week 12 | .94 (.75)

7. Secondary Outcome: Mean Oromandibular Dystonia Quality of Life Questionnaire (OMDQ-25) Score
Description: The OMDQ-25 is a subjective quality of life measurement made for patients with Oromandibular Dystonia. The maximum total score is 100 indicating the highest quality of life. A score of 50 indicates a mediocre quality of life. A lower score indicates perceived lower quality of life.
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport Injections
Number analyzed (Participants) | 18
units on a scale
  Baseline | 47.39 (23.00)
  Week 6 | 43.22 (23.24)
  Week 12: number analyzed (Participants) | 17
  Week 12 | 38.00 (21.42)

8. Secondary Outcome: Mean Global Clinical Impression - Improvement Scale (CGI) Index Score
Description: The Clinical Global Impression - Improvement scale (CGI-I) is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. Responses are scored on a scale from 1 to 7; 1 represents "very much improved" and 7 represents "very much worse".
Time Frame: Week 6, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport Injections
Number analyzed (Participants) | 18
units on a scale
  Week 6 | 2.89 (1.28)
  Week 12: number analyzed (Participants) | 17
  Week 12 | 2.53 (.87)

9. Secondary Outcome: Mean Global Clinical Impression Scale (CGI-S) With Severity Index Score
Description: The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Responses are scored on a scale from 1 to 7; 1 represents "normal, not at all ill" and 7 represents "among the most extremely ill patients".
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Dysport Injections
Number analyzed (Participants) | 18
units on a scale
  Baseline | 4.06 (1.00)
  Week 6 | 3.22 (1.11)
  Week 12: number analyzed (Participants) | 17
  Week 12 | 3.29 (.92)

10. Secondary Outcome: Mean Global Clinical Impression- Efficacy Index Score
Description: The Clinical Global Impression - Efficacy Index is a 4×4 rating scale that assesses the therapeutic effect of treatment. Responses range on a scale from 0 to 4 with 4 being the best response.
Time Frame: Week 6, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport Injections
Number analyzed (Participants) | 18
units on a scale
  Week 6 | 1.51 (.93)
  Week 12: number analyzed (Participants) | 17
  Week 12 | 1.93 (.97)

11. Secondary Outcome: Mean Unified Dystonia Rating Scale (UDRS) Score as Measured by Un-blinded Rater
Description: The UDRS measures dystonia severity. The UDRS is being rated by un-blinded video evaluators regarding severity of subject's dystonia. Scores range from 0 to 10; 0 indicating no dystonia, 5 indicating moderate dystonia, and 10 indicating the worst dystonia.
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport Injections
Number analyzed (Participants) | 18
units on a scale
  Baseline | 4.67 (1.15)
  Week 6 | 3.47 (1.58)
  Week 12: number analyzed (Participants) | 17
  Week 12 | 3.26 (1.47)

12. Secondary Outcome: Mean Global Dystonia Rating Scale Score as Measured by Un-blinded Rater
Description: This scale measures the severity of dystonia for the jaw and tongue by an un-blinded rater. Dystonia is rated from 0 to 10:
  0=No dystonia present, 1=Minimal dystonia, 5=Moderate dystonia,10=Most severe dystonia
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport Injections
Number analyzed (Participants) | 18
units on a scale
  Baseline | 5.67 (1.53)
  Week 6 | 3.94 (2.10)
  Week 12: number analyzed (Participants) | 17
  Week 12 | 3.76 (2.25)

13. Secondary Outcome: Mean Unified Dystonia Rating Scale (UDRS) Score as Measured by Blinded Rater
Description: The UDRS measures dystonia severity. The UDRS is being rated by blinded video evaluators regarding severity of subject's dystonia. Scores range from 0 to 10; 0 indicating no dystonia, 5 indicating moderate dystonia, and 10 indicating the worst dystonia.
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport Injections
Number analyzed (Participants) | 18
units on a scale
  Baseline | 3.50 (1.92)
  Week 6 | 3.47 (1.79)
  Week 12: number analyzed (Participants) | 17
  Week 12 | 3.30 (1.72)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the duration of the study (4 years).
Arm/Group | Dysport Injections
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 9/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport Injections (N=18)
Dysphagia (Gastrointestinal disorders) | 6 (6)
Change in Speech (Nervous system disorders) | 5 (5)
Soft Palate Weakness (Nervous system disorders) | 4 (4)
Xerostomia (Metabolism and nutrition disorders) | 4 (4)
Throat Tightness/Congestion (Gastrointestinal disorders) | 3 (3)
Drooling (Metabolism and nutrition disorders) | 3 (3)
Difficulty Chewing (Metabolism and nutrition disorders) | 2 (2)
Food Falling Out of Mouth (Metabolism and nutrition disorders) | 2 (2)
Coughing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Weight Loss (Investigations) | 2 (2)
Flu-like Symptoms (General disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
The phase 1 study preceding this trial was intended to assess three different Dysport doses. Two participants developed adverse events at the lowest dose in the phase 1 study. Therefore, the lowest dosage level was used for all phase 2 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-03): https://cdn.clinicaltrials.gov/large-docs/70/NCT01921270/Prot_SAP_000.pdf